CLINICAL TRIAL: NCT02058888
Title: Self-controlled Cohort Study of the Amplification and Selection of Antimicrobial Resistance in the Human Intestine
Brief Title: Amplification and Selection of Antimicrobial Resistance in the Intestine
Acronym: ASARI
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Collaborators: University Hospital of Cologne (Other)
Responsible Party: Principal Investigator, Dr. Matthias Willmann, MD, MSc, DTM&H, University Hospital Tuebingen
Other Study IDs: TTU 08.808
Record Dates: First submitted 2014-02-05; First posted 2014-02-10 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Acute Leukaemia
Keywords: metagenomics; antimicrobial resistance; multidrug resistance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bacterial DNA from human stool samples.

SUMMARY:
The worldwide increase in the incidence of multidrug-resistant (MDR) pathogens is alarming. Antimicrobial treatment is a risk factor for the isolation of MDR pathogens and can therefore contribute to the observed trend. Differences in the degree of selection pressure caused by various antimicrobials have not been systematically investigated until today. The aim of the proposed project is the determination of the impact of antibiotic treatment on the copy number of resistance genes in the human intestinal microbiome using metagenome shotgun sequencing. The resistance gene count in the gastrointestinal tract will be determined in a clinical cohorts of patients treated with either ciprofloxacin or cotrimoxazol as monotherapy. The subsequent quantification and comparison of the selection pressure facilitates the application of antibiotics with a lower potential to select for resistance. To achieve this goal, a self-controlled, prospective observational epidemiological study will be performed at two centres of the German Centre for Infection Research (Tübingen, Cologne).

ELIGIBILITY:
Inclusion Criteria:

* male or female patients ≥ 18 years
* patients with acute leukaemia
* admission to one of the 2 study centres
* obtained written consent

Exclusion Criteria:

* treatment with antibiotics in the previous 30 days
* pregnancy
* patients currently treated for HIV and/or hepatitis b/c
* patients who can not estimate scope and consequences of their participation in the study
* patients who will most likely not be able to follow the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be selected from patients admitted to the University Hospital Tuebingen or to the University Hospital Cologne.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Changes from Baseline of Antimicrobial Resistance Gene Content in the human Intestine at three Time Points with respect to different Antibiotic Treatment Regimes. | day 0, day 1, day 3, end of antimicrobial treatment
  Stool samples will be collected from patients at four time points:
  t0 (baseline) The time point serves as a control. The stool sample will be obtained before treatment start.
  t1 (early phase) The time point reflects the early phase at day 1 of treatment with either ciprofloxacin or cotrimoxazol.
  t2 (early-late phase) The time point reflects the early-late phase at day 3 of treatment.
  t3 (late phase) The time point reflects the end of treatment (max. day 7).

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Willmann, MD, Principal Investigator — Institute of Medical Microbiology and Hygiene, Elfriede-Aulhorn-Str.6, 72076 Tuebingen, Germany
Locations (1):
- Institute of Medical Microbiology and Hygiene, University Hospital of Tuebingen, Tübingen, Germany

REFERENCES:
- [Derived] Willmann M, Vehreschild MJGT, Biehl LM, Vogel W, Dorfel D, Hamprecht A, Seifert H, Autenrieth IB, Peter S. Distinct impact of antibiotics on the gut microbiome and resistome: a longitudinal multicenter cohort study. BMC Biol. 2019 Sep 18;17(1):76. doi: 10.1186/s12915-019-0692-y. PMID 31533707